CLINICAL TRIAL: NCT04832581
Title: Effectiveness Of The Self-Care Behavior Development Program For Urinary Tract Infections in Pregnant, Women
Brief Title: Developing Self-care Behaviors for Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esra Çalışkan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECaliskan
Record Dates: First submitted 2021-04-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Urinary Tract Infection During Pregnancy
Keywords: Nursing Care During Pregnancy; Orem Self Care Model; Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: There are two groups in the study, namely the experiment (33) and the control (34) group. The experimental group was included in the program based on the Orem Self Care Model. The program includes anatomical, physiological and hormonal changes during pregnancy, urinary system infections and preventive measures. In the experimental and control groups, the data were collected byface-to-face interview technique and telephone interviews. Pregnant Information Form, Pregnant Evaluation Form, Genital Hygiene Behavior Inventory (GHBI) and routine laboratory testsof pregnant women were used to collect data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group was informed that they participated in a study. After the data collection forms were introduced, written and verbal consents were obtained. Information has been received. The experimental group was included in the program based on the Orem Self Care Model. The program includes anatomical, physiological and hormonal changes during pregnancy, urinary system infections and preventive measures. A phone call was scheduled 2 weeks later. Second evaluation forms were applied. Both groups were informed that the study was concluded.
  Interventions: Behavioral: The Self-Care Behavior Development Program
- Control Group (No Intervention): The control group was informed that they participated in a study. After the data collection forms were introduced, written and verbal consents were obtained. Information has been received. A phone call was scheduled 2 weeks later. Second evaluation forms were applied. After the research was completed, information was given in order to avoid bias and the brochure was delivered. Both groups were informed that the study was concluded.

INTERVENTIONS:
Behavioral: The Self-Care Behavior Development Program — This program, which is based on the Orem Self Care Model, includes anatomical, physiological and hormonal changes, urinary system infections and preventive measures during pregnancy. The program is different from other researches in that it is based on a methodological theory and is created with up-to-date information.
  Arms: Experimental Group

SUMMARY:
The research was designed in a randomized controlled quasi-experimental type in order to reveal the effect of "Self-Care Behaviors Development Program for Urinary Tract Infections" prepared according to Orem's Self Care Model on the behavioral change in pregnant women.

DETAILED DESCRIPTION:
Study Population and Sample The universe of the study consists of all women who have been diagnosed with pregnancy who admitted to the pregnant outpatient clinics of hospitals and who meet the inclusion and exclusion criteria. Pregnant women were selected by simple random sampling method and included in the study.

n=(Nt^2 pq)/(d^2 (N-1)+t^2 pq) According to his formula, n = 29.828625 was found at the significance level of α = 0.05 at 0.05 margin of error.

n = Number of women to be included in the sampling N = the number of participants that make up the universe of the research (3000) p = Frequency of occurrence (0.02) q = frequency of occurrence of the event (1-p) t = t table value at the error level detected at a certain degree of freedom (1.96) d = the desired deviation value (0.05) according to the frequency of occurrence of the event When the urinary system infection is seen as 2% in pregnant women (Ayhan et al.2008) and the number of live births of the hospital in one year is taken as 3000 reference (Hospital archive) α = 0.05 at the significance level of 0.05 The number of pregnant women to be sampled in the margin of error is 30 people. It is planned to work with a total of 60 participants, 30 for the experimental group and 30 for the control group.

Randomization was applied to determine the experimental and control groups. Data Collection Tools Before determining the data collection tools, the literature about the research subject was searched. Tools were determined in accordance with the information obtained from the literature. At the same time, a Self-Care Behaviors Development Program was created, and it was decided to implement the program with the pregnant women in the experimental group by face-to-face meeting and then by phone call. Two forms and an inventory were used to collect data in the study. Data collection tools used in research;

* Pregnant Information Form
* Pregnant Evaluation Form
* Genital Hygiene Behaviors Inventory
* Pregnancy Education Brochure Data Collection The pregnant women who accepted to participate in the study were informed about the purpose and importance of the research, data collection tools and methods, and the flow of the study. While a brochure was given to the pregnant women in the control group (after the end of the study) in the randomization table, the pregnant women in the experimental group were informed that they were included in a training and counseling program and that they would be interviewed again by phone. Each pregnant participating in the study was also informed that she could quit the study at any time.

The data collection of the research took place in 4 stages. Preparation phase Before starting the study, the written permissions of the study (the permission of the ethics committee, the permission of the institution where the study will be conducted and the use of the Genital Hygiene Behavior Inventory used in the study were obtained.

First stage Determination of groups and randomization: It was planned to have an experimental and a control group according to the type of study. Determination of the patients included in the experimental and control groups was made using the randomization program.

Obtaining Informed Volunteer Consent: After obtaining the necessary permissions for the study, the researcher gave written and verbal expressions about the study in a language they understand to the pregnant women who met the inclusion criteria of the study. After the written consent form was signed by the pregnant women who accepted to participate in the study, the study was carried out by the researcher using a face-to-face interview technique.

Second stage After all the necessary permissions and preparations for the study were made, the data collection tools of the study (Pregnant Information Form, Genital Hygiene Behavior Inventory) were filled in in accordance with the information obtained from the patients.

After the information obtained, the "Self-Care Behaviors Development Program for Urinary Tract Infections" prepared for the pregnant women in the experimental group was applied.

Pregnancy Follow-up Form and Genital Hygiene Behavior Inventory were applied to the pregnant women in the experimental group 2 weeks after the end of the program, in order to evaluate the effectiveness of the training by the researcher using the telephone interview technique.

Third stage All information obtained by the researcher and from the patient records were recorded in the Pregnant Information Form, Pregnancy Evaluation Form and Genital Hygiene Behavior Inventory. The recorded data were transferred to the computer environment by the researcher, and the data were evaluated and statistically analyzed.

Data Evaluation The evaluation and statistical analysis of the data were performed in computer environment using the Statistical Pocket Program Statistical Package for the Social Sciences (statistics program for social sciences = SPSS 22.0). In the first stage, percentages and averages were calculated in the calculation of the distribution of the data of the study. In the second stage, when the numerical data met the normal distribution criteria, statistical analysis was performed using an independent sample t test, considering the distribution of normality. Numerical data that did not show normal distribution were evaluated using the Mann Whitney U test. Variables specified in frequency will be analyzed by Chi-square test. P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study,
* To speak and understand Turkish,
* Access to patient records,
* Pregnancy diagnosis by ultrasound

Exclusion Criteria:

* The pregnant woman does not want to participate in the Self-Care Behaviors Development Program for Urinary Tract Infections prepared according to Orem's Self-Care Model,
* Pregnant's use of corticosteroids

Ages: 22 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The research is planned to be conducted with pregnant women.
Enrollment: 67 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Genital Hygiene Behavior Inventory (GHBI) | 2 weeks
  Likert type inventory consisting of 27 questions evaluating genital hygiene behaviors.Inventory was applied to all pregnant women participating in the study at the beginning and at the end of the study.
Pregnant Information Form | 2 weeks
  The form consists of 8 sections including sociodemographic information, information about pregnancy, urinary characteristics, hygiene habits, information about sexuality and pain status, examinations of the pregnant (such as full urinalysis) and the observation form. The form was created by researchers in line with the literature. It was used to take the first anamnesis of the pregnant woman.
Pregnancy Evaluation Form | 2 weeks
  The form consists of six sections including anthropometric information, information about pregnancy, urinary characteristics, hygiene habits, information about sexuality and pain status. The form was created by researchers in line with the literature. It was used for the post-training evaluation of the pregnant woman.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Esra Çalışkan, Istanbul
  - Nevin Hotun Şahin, Istanbul

IPD SHARING:
Plan to Share IPD: No
Research results will be shared.

REFERENCES:
- [Background] Azami M, Jaafari Z, Masoumi M, Shohani M, Badfar G, Mahmudi L, Abbasalizadeh S. The etiology and prevalence of urinary tract infection and asymptomatic bacteriuria in pregnant women in Iran: a systematic review and Meta-analysis. BMC Urol. 2019 May 30;19(1):43. doi: 10.1186/s12894-019-0454-8. PMID 31146773
- [Background] Easter SR, Cantonwine DE, Zera CA, Lim KH, Parry SI, McElrath TF. Urinary tract infection during pregnancy, angiogenic factor profiles, and risk of preeclampsia. Am J Obstet Gynecol. 2016 Mar;214(3):387.e1-7. doi: 10.1016/j.ajog.2015.09.101. Epub 2015 Oct 9. PMID 26450405
- [Result] Amiri FN, Rooshan MH, Ahmady MH, Soliamani MJ. Hygiene practices and sexual activity associated with urinary tract infection in pregnant women. East Mediterr Health J. 2009 Jan-Feb;15(1):104-10. PMID 19469432
- [Result] Emiru T, Beyene G, Tsegaye W, Melaku S. Associated risk factors of urinary tract infection among pregnant women at Felege Hiwot Referral Hospital, Bahir Dar, North West Ethiopia. BMC Res Notes. 2013 Jul 25;6:292. doi: 10.1186/1756-0500-6-292. PMID 23885968
- [Result] Ghouri F, Hollywood A, Ryan K. A systematic review of non-antibiotic measures for the prevention of urinary tract infections in pregnancy. BMC Pregnancy Childbirth. 2018 Apr 13;18(1):99. doi: 10.1186/s12884-018-1732-2. PMID 29653573
- [Result] Haider G, Zehra N, Munir AA, Haider A. Risk factors of urinary tract infection in pregnancy. J Pak Med Assoc. 2010 Mar;60(3):213-6. PMID 20225781
- [Result] Stapleton A, Stamm WE. Prevention of urinary tract infection. Infect Dis Clin North Am. 1997 Sep;11(3):719-33. doi: 10.1016/s0891-5520(05)70382-2. PMID 9378932
- See also: Related Info — http://www.researchgate.net/publication/332443949_Evli_Kadinlarin_Genital_Hijyen_Davranislarinin_Urogenital_Semptomlar_ile_Iliskisi
- See also: Related Info — http://dergipark.org.tr/tr/pub/vansaglik/issue/54113/615967
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/29284
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/29709
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/835961
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/1104822
- See also: Related Info — http://dergipark.org.tr/tr/download/article-file/1039581